CLINICAL TRIAL: NCT05948813
Title: A Phase II Study of TY-9591 Tablets in Patients With EGFR-Mutated Non-small Cell Lung Cancer With Brain Metastases
Brief Title: TY-9591 in the Patients With EGFR Mutations in Advanced NSCLC With Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1601202
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-07

CONDITIONS: NSCLC; EGFR Activating Mutation; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TY-9591 Tablets (Experimental): TY-9591 (160mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: TY-9591
- Osimertinib (Active Comparator): Osimertinib (80mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: TY-9591 — The dose of TY-9591 tablet is 160 mg once daily. A cycle of treatment is defined as 21 days of once daily treatment until meet the of discontinuation criteria.
  Arms: TY-9591 Tablets
Drug: Osimertinib — The dose of Osimertinib is 80 mg once daily. A cycle of treatment is defined as 21 days of once daily treatment until meet the of discontinuation criteria.
  Other Names: Tagrisso
  Arms: Osimertinib

SUMMARY:
This study is to evaluate the efficacy and safety of TY-9591 in first-line treatment of patients with EGFR-sensitive mutation-positive non-small cell lung cancer with brain metastases compared to Osimertinib.

DETAILED DESCRIPTION:
This is an open label, multi-center phase II study to compare the efficacy and safety with Osimertinib in EGFR mutated NSCLC patients with brain metastases. Participants will be randomly assigned to one of the TY-9591 group (160mg orally, once daily) or Osimertinb group (80mg orally, once daily) . Participants can continue to receive study treatment as long as disease progression, meeting criteria for discontinuation of treatment, withdrawal criteria, or study termination (whichever occurred first).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years and <80 years.
2. Patients diagnosed with NSCLC by histology or cytology, with brain metastases.
3. Presence of an activating EGFR-sensitive mutations (including exon 19 deletions, L858R, the above mentioned mutations alone or co-existed with other EGFR-mutated sites).
4. No prior systemic antitumor therapy for locally advanced or metastatic NSCLC.
5. Stable brain metastases that do not require immediate or planned local treatment for it during the study period.
6. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
7. The ECOG score is 0-1, and there is no deterioration 2 weeks before the study, and the expected survival is not less than 3 months.
8. Adequate bone marrow reserve function, and no liver, kidney and coagulation dysfunction.
9. Male patients and female patients of reproductive age should take adequate contraceptive measures from signing informed consent to 3 months after the last study drug treatment; Women of childbearing age have negative pregnancy test results within 7 days of the first dose.
10. Patients having recovered from all grade ≤ 1 toxicities related to previous anticancer therapies (CTCAE v 5.0) except for alopecia, platinum-therapy-related neuropathy (where ≤2 is allowed) before first dose of study treatment.
11. Patients can understand and voluntarily sign the informed consent form.
12. Patient able to comply with study requirements.

Exclusion Criteria:

1. Any of the following treatment:

   1. Previous treatment with EGFR inhibitor;
   2. Previous treatment with Systematic antitumor therapy (including targeted therapy, biotherapy and immunodrug therapy, etc.)；
   3. Previous treatment with standard chemotherapy with 28 days before the first dose of the study drug, and traditional Chinese medicine antitumor therapy within 7 days before the first dose of the study drug;
   4. Previous whole brain radiation therapy (WBRT); Receiving radiation to more than 30% of the bone marrow or with a wide field of radiation that had to be completed within 28 days of the first dose of study treatment; Radiotherapy with a limited field of radiation within 7 days of the first dose of study treatment or palliative radiation therapy for bone metastasis;
   5. Uncontrollable or poorly controlled pleural, abdominal and pericardial effusion;
   6. Uncontrollable cancerous pain; Anesthetic painkillers did not reach a stable dose at the time of enrollment;
   7. Major surgery within 28 days of the first dose of study treatment;
   8. Patients currently receiving (or at least within 14 days prior to receiving the first dose )medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 isoenzyme (CYP)3A4;
   9. Patients who are receiving and need to continue receiving medications during the study that are known to prolong the QTc interval or may cause tachycardia;
   10. Participants in other clinical trials (other than non-interventional clinical trials) within 28 days prior to the first administration of the investigational drug.
2. Patients with primary malignant brain tumors and unstable brain metastases.
3. Patients who have had or have a history of other malignancies within the past 5 years (except cured basal cell or squamous cell carcinoma of the skin, papillary carcinoma of the thyroid gland, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast).
4. The patient had symptoms of spinal cord compression caused by the tumor.
5. Clinically severe gastrointestinal dysfunction may affect the ingestion, transport or absorption of the study drugs.
6. Cardiac function and disease are consistent with the following:

   1. Corrected QT interval(QTc)> 470 milliseconds from 3 electrocardiograms (ECGs);
   2. Any clinically important abnormalities in rhythm;
   3. Any factors that increase the risk of QTc prolongation;
   4. Left ventricular ejection fraction (LVEF) <50%.
7. Active human immunodeficiency virus (HIV), syphilis, hepatitis c virus (HCV) or hepatitis b virus (HBV) infection, with the exception of asymptomatic chronic hepatitis b or hepatitis c carriers.
8. Previous history of interstitial lung disease(ILD) or drug-induced ILD or radiation pneumonitis require steroid treatment, or any evidence of clinically active ILD diseases.
9. Previous allogeneic bone marrow transplant.
10. Pregnant or lactating women.
11. Any other disease or medical condition that is unstable or may affect the safety or study compliance.
12. Hypersensitivity to TY-9591 or similar compounds or excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial Overall Response Rate (iORR) | 36 months
  iORR is defined as the proportion of patients with a best intracranial response of complete response (CR) or partial response (PR) during the study treatment
Intracranial Median Progression Free Survival (iPFS) | 36 months
  iPFS is defined as time from date of first dose of study treatment until the date of first documented intracranial disease progression or death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 36 months
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) during the study treatment
Median Progression Free Survival (PFS) | 36 months
  PFS is defined as time from date of first dose of study treatment until the date of first documented disease progression or death due to any cause
Disease Control Rate (DCR) | 36 months
  DCR is defined as the proportion of patients with a best overall response of complete response (CR) , partial response (PR) or Stable disease (SD) ≥6 weeks during the study treatment
Intracranial Disease Control Rate (iDCR) | 36 months
  iDCR is defined as the proportion of patients with a best intracranial response of complete response (CR) , partial response (PR) or Stable disease (SD) ≥6 weeks during the study treatment
Depth of Response (DepOR) | 36 months
  The Depth of response was defined as the relative change in the sum of the longest diameters of Target lesions (TLs) at the nadir compared to baseline, in the absence of new lesions (NLs) or progression of Non-target lesions (NTLs)
Intracranial Depth of Response (iDepOR) | 36 months
  iDepOR was defined as the relative change in the sum of the longest diameters of intracranial Target lesions (TLs) at the nadir compared to baseline, in the absence of intracranial new lesions (NLs) or progression of intracranial Non-target lesions (NTLs)
Intracranial Time to Response (iTTR) | 36 months
  iTTR is defined as the time from randomization to the first assessment of CR or PR for intracranial tumors
Duration of Response (DoR) | 36 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of first documented disease progression or death due to any cause during the study treatment
Intracranial Duration of Response (iDoR) | 36 months
  iDoR is defined as the time from the date of first documented intracranial response (PR or CR) until the date of first documented disease progression or death due to any cause during the study treatment
Overall Survival (OS) | Up to approximately 60 months
  OS is defined as the time from randomization until death from any cause
Assessment of health-related quality of life (FACT-L) | 36 months
  Change in FACT-L scores relative to Baseline
Safety variables | Up to approximately 60 months
  Adverse events, clinical symptoms, vital signs, ECG's, clinical laboratory safety tests, ect.
Assessment of Karnofsky and NANO | 36 months
  Change in Karnofsky and NANO scores relative to Baseline
Plasma Concentrations of TY-9591 and metabolite | 36 months
  To characterise the pharmacokinetics (PK) of TY-9591 and TY-9591 metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute/Hospital, Chinese Academic of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospitial,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No